CLINICAL TRIAL: NCT04657315
Title: Investigator-initiated and Open-labeled Clinical Trial for Evaluation of Maximum Tolerated Dose, Safety and Efficiency of MSC11FCD Therapy to Recurrent Glioblastoma Patients
Brief Title: Evaluation of Maximum Tolerated Dose, Safety and Efficiency of MSC11FCD Therapy to Recurrent Glioblastoma Patients
Acronym: MSC11FCD-GBM
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CHA University (Other)
Collaborators: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Kyung GI, CHO, Professor, CHA University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHAMC 2019-08-022
Record Dates: First submitted 2020-11-01; First posted 2020-12-08 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Glioblastoma; Adult Gliosarcoma; Neoplasms, Brain; Neoplasms, Germ Cell and Embryonal; Recurrent Glioblastoma
Keywords: Glioblastoma, Mesenchymal stem cells; Brain Tumor; Neoplasms, Germ Cell; Flucytosine; Central Nervous System Neoplasms
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms; Neoplasms, Germ Cell and Embryonal; Central Nervous System Neoplasms | interventions — Cytosine Deaminase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The investigational drug into the Intratumoral administration (Other): The investigational drug in the amount of 1x10^7, 3x10^7cells per dose into the tumor or the tumor removal site using a syringe during surgery
  Interventions: Drug: MSC11FCD

INTERVENTIONS:
Drug: MSC11FCD — Administration period: Single dose Route of administration: Intratumoral administration Dose: 1x10^7, 3x10^7cells/dose Summary: Administer the investigational drug in the amount of 1x107, 3x107cells per dose into the tumor or the tumor removal site using a syringe during surgery.
  Concomitant drug: 5-Flucytosine (prodrug) Dose: 150mg/kg/day
  Directions:
  Administration period and directions: Administer 150m of 5-Flucytosine per kilogram of body weight every 6 hours for a total of 4 times a day (QID) for a duration of 7 days after surgery.
  Route of administration: Oral administration
  Other Names: Mesenchymal stem cells into which the suicide gene, cytosine deaminase (CD)

SUMMARY:
This is a phase I trial evaluating the maximum tolerated dose, safety and efficiency of Mesenchymal stem cells into which the suicide gene, cytosine deaminase (CD), injected into the resection cavity of patients with recurrent glioblastoma.

DETAILED DESCRIPTION:
Not Provided

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 19 to 70
2. Patients diagnosed with recurrent glioblastoma based on medical imaging after receiving standard therapy for glioblastoma
3. Patients scheduled to undergo surgical treatment for recurrent glioblastoma
4. Patients diagnosed with recurrent glioblastoma based on medical imaging (MRI: conventional, diffusion, perfusion, spectroscopy) and confirmed to have tumor cells during surgery based on frozen biopsy
5. Patients whose expected survival period is at least 3 months
6. Patients who have not received any other types of immunotherapy
7. Patients who have been given a sufficient explanation of the purpose and details of the clinical trial and the characteristics of the investigational drug from an investigator and who signed the consent form or had a legal guardian or representative sign the consent form prior to the beginning of this clinical trial
8. Patients who have waited for at least four weeks after treatment using cytotoxic drugs in order to eliminate the possibility of impact and effects from other therapeutic agents (23 days after the last administration in case of undergoing standard therapy using temozolomide)

Exclusion Criteria:

1. Patients who have primary glioblastoma
2. Patients with dihydropyrimidine dehydrogenase (DPD) deficiency
3. Patients who cannot undergo a contrast (gadolinium) enhanced MRI scan due to a certain condition (pacemaker, etc.) or cannot undergo an MRI scan according to the clinical trial schedule due to any other reasons
4. Patients to whom Gliadel water was applied during surgery
5. Patients who are deemed to have a serious dysfunction in any of the major organs (liver, kidneys, bone marrow, lungs, heart) by the investigator
6. Patents who have other types of malignant tumor aside from glioblastoma or who have had malignant tumor in the past 5 years
7. Patients who uncontrolled hypotension or hypertension
8. Diabetic patients who are currently receiving insulin therapy or who need insulin therapy
9. Patients who are deemed to have a serious infectious disease by the investigator: sepsis, hepatitis A, hepatitis B or hepatitis C (in the case of hepatitis B and C viruses, however, carriers may be enrolled at the investigator's discretion) or tested positive in a serological test for the human immunodeficiency virus (HIV)
10. Karnofsky Performance Scale < 60
11. Patients with an autoimmune disease affecting the central nervous system (multiple sclerosis, myasthenia gravis, acute disseminated encephalomyelitis, etc.)
12. Patients with a history of allergic reactions to flucytosine (5-FC) and/or its excipients or 5-fluorouracil (5-FU)
13. Pregnant or lactating women or patients who plan on getting pregnant during the clinical trial or refuses to choose an appropriate method of contraception
14. Patients who have participated in a different clinical trial no more than 30 days prior to registering for this clinical trial
15. Patients who are deemed to be unfit for this clinical trial by the investigator

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | after treatment discontinuation for approximately 1 years
  Assessment of the maximum tolerated dose based on the 3+3 method
  * Blood concentrations of 5-FC and 5-FU(Day 1, Day 3, Day 7)
  * MSC11FCD concentrations (MSCCD detection) (Day 0, 3months, 6months, 12months)
Number Of Adverse Events related to the treatment | Baseline, Day0, 1 month, 3 months, 6 months, 12 months
  Evaluate the number of adverse event related to the treatment according to CTCAE V4.0 during the trial (including clinically significant changes in physical examination, radiographic images, safety lab tests, vital signs)

SECONDARY OUTCOMES:
Overall Survival improvement (OS) | Study entry through the end of the study, up to 12 months
  OS is defined as the time from the date of MSC injection to the date of death due to any cause.
Progression Free Survival (PFS) | Study entry through the end of the study, up to 12 months
  The progress-free survival analysis shall be based on the RANO criteria.
Tumor assessment in regard to the investigational drug based on the RANO criteria | At Baseline, 1month, 3months, 6months, 12months
  Assess the treatment groups participating in this clinical trial based on the RANO criteria.
  Compare and present the disease control rates by calculating the ratio of the number of subjects responding to treatment (complete response: CR, partial response: PR, stable disease: SD) among the treatment groups and control group assessed based on the RANO criteria.
Clinical efficacy assessment | At Baseline, 1month, 3months, 6months, 12months
  Karnofsky performance status (KPS) assessment

CONTACTS AND LOCATIONS:
Overall Officials: Kyunggi Cho, MD,PhD, Principal Investigator — CHA University
Locations (1):
- Bundang CHA Medical Center, Seongnam, Kyunggido, South Korea

IPD SHARING:
Plan to Share IPD: No